CLINICAL TRIAL: NCT03300284
Title: Decision Making and Psychological Outcomes in Low-Risk Papillary Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-382
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Thyroid Cancer
Keywords: Quality of Life; Decision Making; 17-382
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thyroid cancer: This study does not involve any intervention, but rather data collection on patient and physician preferences and beliefs, communication, and patient psychological outcomes.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Quality of Life Questionnaires

SUMMARY:
This study is being done to understand the decision-making process regarding management choice in low-risk papillary thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, write, and communicate in English Patients who have been diagnosed with LR-PTC as described above
* For Aim 1, adults with recently diagnosed LR-PTC who have not yet made a choice between surgery and AS
* For Aim 2, adults with LR-PTC who made a decision about surgery or AS at least 3 months prior, but no more than 4 years prior to their routine follow-up visit at which they are being recruited for this study.
* Active patients of MSK and participating institutions

Exclusion Criteria:

* Patients who have been diagnosed with a tumor greater than 2 cm
* Patients with clinically suspicious lymphadenopathy in the neck
* Patients with evidence of gross ETE after a biopsy of the papillary thyroid tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted primarily in the MSK endocrinology and surgery clinics, which have a large volume of patients with LR-PTC choosing both surgery and AS. We also expect to expand this study to several clinics within the MSK Alliance Network and outside participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
influencing decision making pre-visit | 3 years
  Patients will complete a pre-visit questionnaire and the patient-physician interaction during the visit will be recorded and subjected to qualitative analysis for extraction of variables representing the presence of elements of shared decision making and strength of physician influence.
influencing decision making post-visit | 3 years
  Patients will complete a post-visit questionnaire, and the patient-physician interaction during the visit will be recorded and subjected to qualitative analysis for extraction of variables representing the presence of elements of shared decision making and strength of physician influence.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Roman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Hartford Healthcare (Data Collection), Hartford, Connecticut
  - Memorial Sloan Kettering Monmouth (Consent and Follow up), Middletown, New Jersey
  - MAIMONIDES MEDICAL CENTER (Data collection only), Brooklyn, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm